CLINICAL TRIAL: NCT05896007
Title: Zanubrutinib Combined With Rituximab and Chemotherapy for Newly-Diagnosed Primary Central Nervous System Large B-Cell Lymphoma Patients Intolerant to Haematopoietic Stem Cell Transplantation
Brief Title: Zanubrutinib Combined With Rituximab and Chemotherapy for Newly-Diagnosed PCNSLBCL Patients Intolerant to HSCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zana
Record Dates: First submitted 2023-05-01; First posted 2023-06-09 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: PCNSL
Keywords: PCNSL; zanubrutinib
MeSH Terms: interventions — zanubrutinib; Rituximab; Methotrexate; Temozolomide

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ZR-chemo (Experimental): Drug: Zanubrutinib, Rituximab and MTX (or TMZ, if intolerant to MTX)
  Interventions: Drug: Zanubrutinib; Drug: Rituximab; Drug: Methotrexate; Drug: Temozolomide

INTERVENTIONS:
Drug: Zanubrutinib — 160 mg bid po, until disease progression, intolerance of drug toxicity or death, otherwise maintaining during the 1st year in 2 years of follow-up
  Other Names: brukisa
Drug: Rituximab — 375 mg/m^2 ivgtt, D0 of each 28-day cycle
Drug: Methotrexate — 3.5 g/m^2 ivgtt, D1 of each 28-day cycle
Drug: Temozolomide — 150 mg/m^2 ivgtt, D1-D5 of each 28-day cycle

SUMMARY:
This single-center, open, single-arm study aim to evaluate the efficacy and tolerability of a therapy introducing zanubrutinib on the basis of rituximab and methotrexate (MTX) [or temozolomide (TMZ), if intolerant to MTX] in treating patients newly diagnosed with primary CNS large B-cell lymphoma and intolerant to HSCT.

DETAILED DESCRIPTION:
Participants will receive zanubrutinib in addition to first-line therapy consisting of rituximab and either MTX or TMZ. After treatment of 6 cycles with the new regimen, the patients achieving CR or PR would go on to receive zanubrutinib maintenance of 1 year (if tolerable).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old;
* Histopathologically confirmed CD20 positive primary large B-cell lymphoma of the central nervous system (CNS) or primary vitreoretinal lymphoma according to the 5th edition of the World Health Organization (WHO) Classification of Haematolymphoid Tumours [primary large B-cell lymphoma of the CNS previously named as primary diffuse large B-cell lymphoma (DLBCL) of the CNS in the revised 4th edition];
* Life expectancy of > 3 months (in the opinion of the investigator);
* Creatinine Clearance Rate (CCR) ≥ 50 mL/min or estimated Glomerular Filtration Rate (eGFR) ≥ 60 mL/(min·1.73 m^2);
* International Normalized Ratio (INR) ≤ 1.5 and activated Partial Thromboplastin Time (aPTT) ≤ 1.5 times the upper limit of normal;
* Left Ventricular Ejection Fraction (LVEF) ≥ 50%;
* Agreeing to provide written informed consent prior to any special examination or procedure for the research on their own or legal representative.

Exclusion Criteria:

* Pregnant or lactating women;
* Known Hepatitis B Virus (HBV) and/or Hepatitis C Virus (HCV) infection (HBV infection refers to HBV-DNA > detectable limit);
* With acquired or congenital immunodeficiency;
* With congestive heart failure in 6 months before enrollment, New York Heart Association (NYHA) heart function class III or IV, or LVEF < 50%;
* Known to be allergic to the test drug ingredients;
* Diagnosed with or being treated for malignancy other than lymphoma;
* With severe infection;
* Substance abuse, medical, psychological, or social conditions that may interfere with the subjects' participation in the study or evaluation of the study results;
* Deemed unsuitable for the group.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year Progression-Free Survival | 2 years
  Progression-free survival was defined as the time from the date of first treatment until the date of the first documented day of disease progression or relapse, according to 2014 Lugano criteria, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Baseline up to data cut-off (up to approximately 2 years)
  The ORR is defined as percentage of participants with overall response including complete response (CR), unconfirmed complete response (CRu) and partial response (PR), on the basis of investigator assessments, according to the 2005 Response Criteria of the International Primary CNS Lymphoma Collaborative Group (IPCG).
Complete Response (CR) Rate | Baseline up to data cut-off (up to approximately 2 years)
  The CR rate is defined as the proportion of patients with CR/CRu according to the 2005 Response Criteria of the International Primary CNS Lymphoma Collaborative Group (IPCG).
Overall Survival (OS) | Baseline up to data cut-off (up to approximately 2 years)
  Overall survival is defined as the time from the date of first treatment to the date of death from any cause.
Adverse Events | Baseline up to data cut-off (up to approximately 2 years)
  Any harmful reaction that occurs during the treatment of a disease according to the normal usage and dosage of a drug, which is unrelated to the purpose of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No